CLINICAL TRIAL: NCT01778712
Title: Developing an Intervention to Prevent Visceral Adipose Tissue Accumulation in Premenopausal Women: WISHfit Phase 2
Brief Title: Developing an Intervention to Prevent Visceral Adipose Tissue Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lynda Powell, PhD, MEd, PhD, MEd, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09090108; 5U01HL097894-03 (NIH)
Record Dates: First submitted 2012-10-24; First posted 2013-01-29 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Menopause; Visceral Adipose Tissue Accumulation; Abdominal Obesity; Obesity; Overweight
Keywords: Multi-level intervention; Menopause; Body composition; Abdominal adipose tissue; Visceral adipose tissue; Perceived stress; Computed tomography; Dual energy X-ray absorptiometry
MeSH Terms: conditions — Obesity, Abdominal; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Multi-level intervention
  Interventions: Behavioral: Multi-level intervention

INTERVENTIONS:
Behavioral: Multi-level intervention — The development of a lifestyle program intended to intervene on the individual, social network and community over two years
  Other Names: Lifestyle program

SUMMARY:
The aim of this study is to develop an intervention that will produce a sustained improvement in physical activity and chronic stress as a means to slow the menopause-related accumulation of visceral adipose tissue in mid-life women.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Beverly or Morgan Park neighborhood of Chicago or contiguous neighborhoods
* Female
* African American or Caucasian
* Age 42 years or older
* Intact uterus, at least one functioning ovary, at least one menstrual period in the last 12 months prior to screening.
* Sufficient motivation level to make lifestyle changes, as determined by WISHFIT staff.

Exclusion Criteria:

* Hysterectomy
* Physical activity > 90 min per week
* Metabolic conditions or use of medications that affect weight of visceral adipose tissue (diabetes, acquired immune deficiency syndrome, weight > 300 lbs)
* Presence or history of major psychiatric comorbidity (i.e. dementia, schizophrenia, bipolar disorder, alcohol/drug addiction) in the last 6 months
* History of inpatient mental health treatment
* Currently prescribed antipsychotic medication
* History of hallucinations or bizarre thoughts
* Current pregnancy
* Has been told by a physician that it is unsafe to engage in physical activity
* An illness expected to limit functional status or life expectancy, including: heart failure, recent heart attack, liver cirrhosis, kidney failure, oncologic conditions, history or heart surgery, angioplasty or artery stenting.

Min Age: 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in visceral adipose tissue, as measured by CT | At two years from baseline
  <4% gain in visceral adipose tissue over a 2-year period

SECONDARY OUTCOMES:
Effects of the multi-level intervention | At two years from baseline
  Physical activity as assessed by accelerometer (min/week of >= 3 MET)
Effects of the multi-level intervention | At two years from baseline
  Proportion or participants meeting a 120 min/week physical activity goal
Effects of the multi-level intervention | At two years from baseline
  Vitality subscale of the SF36 questionnaire
Effects of the multi-level intervention | At two years from baseline
  Assess Dietary changes (vegetable, protein, fat, sugar-sweetened beverage consumption)
Effects of the multi-level intervention | At two years from baseline
  Assess Perceived stress
Effects of the multi-level intervention | At two years from baseline
  Assess Perceived social support
Effects of the multi-level intervention | At two years from baseline
  Knowledge of menopausal effects on health in the target community, as assessed by the "man on the street" survey

OTHER OUTCOMES:
Change in body composition | At two years from baseline
  * Change in waist girth and BMI
  * Subcutaneous and visceral adipose tissue as measured by CT
  * Body composition as measured by dual energy X-ray absorptiometry (fat, lean mass)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda H. Powell, PhD, MEd, Principal Investigator — Rush University Medical Center
Locations (1):
- Department of Preventive Medicine, Rush University Medical Center, Chicago, Illinois, United States